CLINICAL TRIAL: NCT07192770
Title: Prospective Observational Evaluation of Supportive Care Strategies for G-CSF-Induced Bone Pain and Associated Symptoms in Patients With Solid Tumors
Brief Title: G-CSF-Induced Bone Pain and Supportive Care Approaches
Acronym: GCSF-PAIN
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncology Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-196; AEŞH-EK-2025-196 (Other: Ankara Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors; Chemotherapy-induced Neutropenia
Keywords: G-CSF; Bone Pain; Chemotherapy Supportive Care; Quality of Life; Fatigue; Depression; Sleep Quality; Patient-Reported Outcomes; G-CSF-Induced Bone Pain
MeSH Terms: conditions — Fatigue; Depression; Sleep Initiation and Maintenance Disorders | interventions — Granulocyte Colony-Stimulating Factor; pegfilgrastim; Filgrastim; Palliative Care; Analgesics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Receiving G-CSF During Chemotherapy: Adult patients (aged 18-70 years) with histologically or cytologically confirmed solid tumors who are receiving chemotherapy with prophylactic G-CSF (granulocyte colony-stimulating factor). Patients are consecutively enrolled and assessed for bone pain and supportive care needs before and one week after G-CSF administration.
  Interventions: Biological: Granulocyte colony-stimulating factor (G-CSF); Other: Supportive Care (Analgesic and Non-Pharmacological Strategies)

INTERVENTIONS:
Biological: Granulocyte colony-stimulating factor (G-CSF) — Patients receive chemotherapy with prophylactic G-CSF (granulocyte colony-stimulating factor) as part of routine clinical care. Both short-acting (filgrastim) and long-acting formulations (pegfilgrastim, lipegfilgrastim) may be used according to standard oncology practice. The study does not assign the intervention but observes supportive care strategies and patient-reported outcomes related to G-CSF-induced bone pain.
  Other Names: Lipegfilgrastim; Filgrastim; Pegfilgrastim
Other: Supportive Care (Analgesic and Non-Pharmacological Strategies) — Supportive care strategies including analgesic use (NSAIDs, opioids, antihistamines) and non-pharmacological interventions (rest, exercise, local heat/cold, relaxation techniques) will be recorded as part of routine practice. The study does not randomize or assign supportive care but documents their use and association with bone pain outcomes.
  Other Names: Non-drug supportive measures; Analgesics

SUMMARY:
This prospective observational study aims to evaluate bone pain and related symptoms in patients with solid tumors receiving granulocyte colony-stimulating factor (G-CSF) during chemotherapy. A total of 128 patients will be enrolled at Ankara Etlik City Hospital. Pain severity will be assessed using the Visual Analog Scale (VAS), and supportive care strategies such as analgesics and non-pharmacological approaches will be documented. Patient-reported outcomes, including quality of life, fatigue, anxiety, depression, and sleep quality, will also be evaluated before and one week after G-CSF administration. The findings are expected to provide practical insights into the management of G-CSF-induced bone pain and improve supportive care practices.

DETAILED DESCRIPTION:
Granulocyte colony-stimulating factor (G-CSF) is widely used for primary or secondary prophylaxis of chemotherapy-induced neutropenia. Despite its clinical benefits, G-CSF frequently induces bone pain, which negatively affects treatment adherence, quality of life, and overall patient comfort. This prospective observational study is designed to systematically evaluate bone pain, quality of life, functional status, mood, and sleep quality in patients with solid tumors receiving G-CSF. A total of 128 participants will be consecutively enrolled at Ankara Etlik City Hospital.

Study Cohort:

All enrolled patients will be adults (aged 18-70 years) with histologically or cytologically confirmed solid tumors receiving chemotherapy with prophylactic G-CSF (filgrastim, pegfilgrastim, or lipegfilgrastim). Participants will be consecutively recruited and assessed for bone pain and supportive care needs before and one week after G-CSF administration. If different G-CSF agents are used, subgroup analyses will be performed according to the type of G-CSF received.

Study Design and Visits:

Eligible patients will be assessed at baseline (before G-CSF administration) and one week after G-CSF. Data will include demographic and clinical characteristics, treatment details, laboratory parameters, and patient-reported outcomes. Pain intensity will be measured using the Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst possible pain). A ≥20% reduction will be considered a clinically meaningful improvement.

Patient-Reported Outcomes and Validation:

EORTC QLQ-C30 (Quality of Life Questionnaire-Core 30): Validated in Turkish cancer populations. Scores range from 0-100; higher functional and global health scores indicate better outcomes, whereas higher symptom scores reflect greater symptom burden.

FACT-G (Functional Assessment of Cancer Therapy-General): Turkish validation is available. Scores range from 0-108; higher scores indicate better overall quality of life.

FACT-F (Fatigue Subscale): Part of the FACT measurement system, validated in Turkish cancer patients. Scores range from 0-52; higher scores indicate lower fatigue severity.

PHQ-9 (Patient Health Questionnaire-9): Turkish validation established. Scores range from 0-27. Cut-offs: 5-9 mild, 10-14 moderate, 15-19 moderately severe, ≥20 severe depression.

GAD-7 (Generalized Anxiety Disorder-7): Validated in Turkish. Scores range from 0-21. Cut-offs: 5 mild, 10 moderate, ≥15 severe anxiety.

Beck Depression Inventory (BDI): Validated Turkish version used. Scores range 0-63. Cut-offs: 0-9 minimal, 10-18 mild, 19-29 moderate, 30-63 severe depression.

PSQI (Pittsburgh Sleep Quality Index): Turkish validation established. Global scores range from 0-21; scores >5 indicate poor sleep quality.

Study Outcomes:

The primary outcome is the change in VAS bone pain scores from baseline to one week after G-CSF administration. Secondary outcomes include changes in QLQ-C30, FACT-G, FACT-F, PHQ-9, GAD-7, BDI, and PSQI scores. Analgesic use and correlations between demographic/clinical features (age, ECOG status, tumor type) and supportive care strategies will also be explored.

Significance:

This study is expected to generate real-world evidence on the prevalence, severity, and management of G-CSF-induced bone pain in patients with solid tumors. Incorporating validated patient-reported outcome tools with established cut-offs ensures methodological rigor and facilitates cross-study comparability. Results may guide clinicians in selecting effective supportive interventions, reduce symptom burden, and improve adherence to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Histologically or cytologically confirmed solid tumor
* Receiving chemotherapy with prophylactic or secondary prophylactic G-CSF (filgrastim, pegfilgrastim, or lipegfilgrastim)
* ECOG performance status 0-3
* Able to complete patient-reported outcome questionnaires (VAS, QLQ-C30, FACT-G, FACT-F, PHQ-9, GAD-7, BDI, PSQI)
* Written informed consent provided

Exclusion Criteria:

* Known bone metastases (confounds bone pain assessment)
* Use of NSAIDs, opioids, or antihistamines within 48 hours prior to G-CSF administration
* Patients not indicated for G-CSF prophylaxis
* Severe cognitive impairment or communication barrier preventing completion of questionnaires
* Active concurrent malignancy requiring systemic therapy
* Known hypersensitivity to G-CSF or supportive care medications
* Investigator judgment that participation may compromise data integrity or patient safety
* ECOG performance status 4

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients (aged 18-70 years) with histologically or cytologically confirmed solid tumors, receiving chemotherapy and prophylactic G-CSF at Ankara Etlik City Hospital. Participants will be consecutively recruited, without randomization, as part of routine clinical care. The study population represents a real-world oncology cohort, designed to capture the prevalence, severity, and management of G-CSF-induced bone pain and related quality-of-life outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-09-27 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Bone Pain Score (0-10) | Baseline and 1 week after G-CSF administration
  Patient-reported bone pain intensity using the Visual Analog Scale (VAS, range 0-10; 0 = no pain, 10 = worst pain). A ≥20% reduction in score is considered a clinically meaningful improvement.

SECONDARY OUTCOMES:
Change in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health/Quality of Life Score (0-100) | Baseline and 1 week after G-CSF administration
  Change in global health status/quality of life score from the EORTC QLQ-C30 (0-100 scale). Higher scores indicate better quality of life. Turkish validation available.
Change in Functional Assessment of Cancer Therapy-General (FACT-G) Total Score (0-108) | Baseline and 1 week after G-CSF administration
  Change in FACT-G total score (0-108). Higher scores indicate better overall quality of life. Turkish validation available.
Change in Functional Assessment of Cancer Therapy-Fatigue (FACT-F) Subscale Score (0-52) | Baseline and 1 week after G-CSF administration
  Change in FACT-F subscale score (0-52). Higher scores indicate less fatigue. Turkish validation available.
Change in Patient Health Questionnaire-9 (PHQ-9) Depression Score (0-27) | Baseline and 1 week after G-CSF administration
  Change in PHQ-9 depression score (0-27). Cut-offs: 5-9 mild, 10-14 moderate, 15-19 moderately severe, ≥20 severe depression. Turkish validation available.
Change in Generalized Anxiety Disorder-7 (GAD-7) Score (0-21) | Baseline and 1 week after G-CSF administration
  Change in GAD-7 anxiety score (0-21). Cut-offs: 5 mild, 10 moderate, ≥15 severe anxiety. Turkish validation available.
Change in Beck Depression Inventory (BDI) Score (0-63) | Baseline and 1 week after G-CSF administration
  Change in BDI score (0-63). Cut-offs: 0-9 minimal, 10-18 mild, 19-29 moderate, 30-63 severe depression. Turkish validation available.
Change in Pittsburgh Sleep Quality Index (PSQI) Score (0-21) | Baseline and 1 week after G-CSF administration
  Change in PSQI global score (0-21). Higher scores indicate poorer sleep quality. A global score >5 indicates poor sleep. Turkish validation available.
Analgesic Use During Study Period (%) | Baseline to 1 week after G-CSF administration
  Type and frequency of analgesics (NSAIDs, opioids, antihistamines) and non-pharmacological supportive measures recorded during follow-up.

OTHER OUTCOMES:
Correlation Between Change in Visual Analog Scale (VAS, 0-10) Bone Pain Score and Supportive Care Strategy | Baseline to 1 week after G-CSF administration
  Exploratory correlation of supportive care type (NSAIDs, opioids, antihistamines, non-pharmacological measures) with change in VAS pain score.
Correlation Between Change in Visual Analog Scale (VAS, 0-10) Bone Pain Score and G-CSF Formulation | Baseline to 1 week after G-CSF administration
  Exploratory correlation of change in VAS pain score according to G-CSF formulation used (filgrastim, pegfilgrastim, lipegfilgrastim).
Correlation Between Change in Visual Analog Scale (VAS, 0-10) Bone Pain Score and Baseline Demographic/Clinical Factors | Baseline to 1 week after G-CSF administration
  Correlation of change in VAS pain score with baseline factors (age, sex, ECOG performance status, tumor type).
Correlation Between Change in Visual Analog Scale (VAS, 0-10) Bone Pain Score and Change in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Score (0-100) | Baseline to 1 week after G-CSF administration
  Correlation analysis between change in VAS pain score and change in EORTC QLQ-C30 global health/quality-of-life score.
Correlation Between Change in Visual Analog Scale (VAS, 0-10) Bone Pain Score and Change in Functional Assessment of Cancer Therapy-General (FACT-G) and Functional Assessment of Cancer Therapy-Fatigue (FACT-F) Scores | Baseline to 1 week after G-CSF administration
  Correlation analysis between change in VAS pain score and change in FACT-G total (0-108) and FACT-F fatigue subscale (0-52).
Correlation Between Change in Visual Analog Scale (VAS, 0-10) Bone Pain Score and Change in Pittsburgh Sleep Quality Index (PSQI) Global Score (0-21) | Baseline to 1 week after G-CSF administration
  Correlation between change in VAS pain score and change in PSQI global score (0-21; >5 indicates poor sleep quality).
Predictors of Clinically Meaningful Pain Improvement (≥20% Reduction in Visual Analog Scale [VAS] Score) | Baseline to 1 week after G-CSF administration
  Multivariable logistic regression to identify predictors of ≥20% reduction in VAS pain score (Yes/No) at 1 week, including supportive care type, G-CSF formulation, and baseline characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Enes Yeşilbaş, MD, Principal Investigator — Etlik City Hospital Medical Oncology Department
Locations (1):
- Etlik City Hospital Medical Oncology Department, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No